

# Prevention of Eating Habits Associated with Obesity in Adolescents through a Wise Intervention

**Informed Consent** 

February 21, 2023



#### **FACULTY OF HEALTH SCIENCES UNIVERSITY OF DEUSTO**

Avenue of the Universities, 24 48007 Bilbao, Vizcaya

This consent form provides information about a research project being conducted at your child's school in collaboration with the University of Deusto that aims to evaluate the effectiveness of brief smart interventions aimed at **preventing obesity in adolescence.** 

Below, you will find all relevant information regarding the project. Once you have read the information, if you do **NOT** want your child to participate in this project, please complete the consent form and return it to your child's school **within 3 days.** If you consent to your child's participation, you **do not need** to complete the form or return it.

## 1. Purpose of the Project:

The main objective of the intervention will be to reduce the intake of unhealthy foods and increase the intake of healthy foods in adolescents, in order to prevent adolescent obesity.

The intervention takes place in a single session of approximately 60 minutes duration. Two intervention formats are used, randomly assigning participants to classrooms. Subsequently, all participants can receive the intervention that was not delivered, provided it is proven to be effective.

The interventions consist of exercises such as: reading materials related to eating habits and stories from other students. In addition, they will engage in writing and/or interactive activities. All students in your child's class have been invited to participate.

## 2. What will my child be required to do?

If you allow your child to participate in this study, you will be asked to:

- Participate in the intervention lasting 60 minutes.
- Complete a 10-20 minute questionnaire the very same day of the intervention and one week and three months after the intervention.

# 3. How will researchers protect the privacy of participants?

This study has the approval of the Research Ethics Committee of the University of Deusto. The researchers will protect the privacy of all participants. No names or surnames will be indicated anywhere. Assessment and intervention data will be linked by a code known only to the participant.

# 4. How will the researchers share the results of the project?

Your child's school will receive a final report reflecting the results of the program evaluation that may be distributed to all parents.

#### 5. Are there any risks or benefits for my child?

There are no foreseeable risks associated with participating in this project. The

intervention and questionnaires are regular school activities. The intervention may be beneficial for a high percentage of students.

## 6. Does my child have to participate?

Consent is optional. Your decision whether or not to allow your child to participate will not affect your current or future relationship with the University of Deusto, the school or your child's teacher. If you decide to allow your child to participate, he/she will be asked if he/she agrees to participate and if your child agrees, he/she will receive all necessary instructions. In addition, he/she is free to stop participating at any time without penalty or adverse consequence. You may also initially allow your child to participate in the study and then change your mind without penalty. This research study will be conducted during regular classroom activities. However, if you do not want your child to participate, a different activity will be available for him/her. Your child will be offered the opportunity to use his/her time to read or do homework.

### 7. What will happen if my child doesn't want to participate?

In addition to your permission, your child must agree to participate in the study. If he/she does not wish to participate, he/she will not be included in the study and there will be no penalty. Even if he/she initially agrees to participate in the study, he/she can change his/her mind later without penalty.

## 8. Will there be any compensation?

There will be no monetary compensation for participation. However, at the end of the study gift vouchers will be raffled in each class. These gift vouchers can be exchanged in a department store.

#### 9. Who has reviewed the study?

The project has been reviewed by the Ethics Committee of the University of Deusto and by the school principals. The school will not carry out the project activities. The study will be carried out by researchers from the University of Deusto.

## 10. Who can I contact with in case I have questions about the study?

- Ainara Echezarraga (telephone: 944139000 (ext. 2147); email: a.echezarraga@deusto.es)
- Nerea Cortazar (telephone: 944139000 (ext. 2668); email: nerea.cortazar@deusto.es)
- Liria Fernández (telephone: 944 139 000 (ext. 2800); email: liria.fernandez@deusto.es)
- Izaskun Orue (telephone: 944139000) (ext. 2935); email: izaskun.orue@deusto.es)
- Esther Calvete (telephone: 944139000 (ext. 2847); email: esther.calvete@deusto.es)

| This page should <b>ONLY</b> be signed if you <b>DON'T</b> want your child to participate in this project. |
|---|
| Your signature indicates that you have read the information above and have decided <b>NOT to allow</b> you child to participate in this project. |
| If you give your permission for your child to participate, you do not have to complete this form. |
| □ <b>NO</b> , my child <b>CAN'T</b> participate in this project. |
| Name and Surname of the Student |
| Name and Sumame of the Student |
| Parent or Guardian's Signature Date: |